CLINICAL TRIAL: NCT04183881
Title: An Extension Study of Brodalumab in Subjects With Plaque Psoriasis (Psoriasis Vulgaris, Psoriatic Arthritis), Pustular Psoriasis (Generalized) and Psoriatic Erythroderma
Brief Title: A Phase 4 Clinical Study of Brodalumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4827-005 (post market)
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis; Pustular; Psoriasis, Palmaris Et Plantaris; Psoriatic Erythroderma
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brodalumab 210mg SC (Experimental): Brodalumab 210mg subcutaneous injection
  Interventions: Drug: Brodalumab 210mg SC

INTERVENTIONS:
Drug: Brodalumab 210mg SC — 210 mg, subcutaneous dosing, every 2 weeks

SUMMARY:
This study [4827-005 (post market)] is designed to evaluate the safety and efficacy of long-term exposure to brodalumab in subjects with plaque psoriasis (psoriasis vulgaris, psoriatic arthritis) who have completed Study 4827-003 (Study 003) and in subjects with pustular psoriasis (generalized) or psoriatic erythroderma who have completed the Study 4827-004 (Study 004). 4827-005 study was conducted as phase 3 clinical trial until July 4th 2016 (approval date in Japan). After that date 4827-005 study was switched to phase 4 study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed the written informed consent form to participate in this study
* Subject has completed the study 4827-005 (phase 3)

Exclusion Criteria:

* Subject has had a serious infection, defined as requiring systemic treatment with antibiotics or antivirals (excluding oral administration)
* Subject has been judged to be ineligible for participation in the study by the investigators/sub investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Incidence and types of adverse events and adverse reactions | 28 weeks
Anti-KHK4827 antibody | 28 weeks

SECONDARY OUTCOMES:
Change in psoriasis area and severity index (PASI) compared to the data obtained before the first dose of investigational product in this study. | 28 weeks
Percent improvement in PASI | 28 weeks
PASI 50, 75, 90, and 100 | 28 weeks
Static physician's global assessment (sPGA) of "0 (clear) or 1(almost clear)" | 28 weeks
sPGA of "0 (clear)" | 28 weeks
Change in body surface area involvement (BSA) of lesion | 28 weeks
Clinical Global Impression (CGI) | 28 weeks
American College of Rheumatology (ACR) 20 | 28 weeks
Pustular symptom score | 28 weeks
  This score indicate the severity of generalized pustular psoriasis (GPP). The severity of GPP (0:none-3:severe) is classified as mild(1), moderateor(2) severe(3) based on a total score after rating skin symptoms (erythema, pustules and edema) and systemic inflammation accom-panied by certain laboratory findings (fever, white blood cellcount, and serum CRP and albumin levels).
Serum KHK4827 concentration | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Jikei University Scoole of Medicine, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided